CLINICAL TRIAL: NCT07166276
Title: Association of Coffee Consumption With Periodontal Health and Disease: An Observational Study
Brief Title: Association of Coffee With Periodontal Status
Acronym: acpc
Status: Completed | Type: Observational
Sponsor: Tuğba ŞAHİN (Other)
Responsible Party: Sponsor-Investigator, Tuğba ŞAHİN, Assistant professor, Abant Izzet Baysal University
Organization: Abant Izzet Baysal University (Other)
Other Study IDs: 2024/311
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Periodontal Diseases
Keywords: coffee; periodontal disease; periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — Coffee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Periodontitis: It refers to a chronic inflammatory disease of the supporting tissues of the teeth, characterized by progressive destruction of the periodontal ligament and alveolar bone, with pocket formation and/or gingival recession.
  Interventions: Other: coffee
- Gingivitis: It refers to a reversible inflammation of the gingival tissues without loss of periodontal attachment. The condition is primarily induced by dental plaque accumulation and is characterized clinically by signs such as gingival redness, swelling, and bleeding on probing.
  Interventions: Other: coffee
- Periodontal health: Periodontal health refers to the absence of clinical signs of inflammation in the periodontium, with stable supporting tissues and no evidence of attachment loss or bone destruction.
  Interventions: Other: coffee

INTERVENTIONS:
Other: coffee — The type of coffee consumed, the daily amount of coffee, and the frequency of consumption were measured.

SUMMARY:
A total of 318 patients applying to Bolu Abant İzzet Baysal University will be included in the study. Based on anamnesis, radiographic examination, and the 2018 classification of periodontal diseases, the participants will be categorized into three groups: periodontal health (n=106), gingivitis (n=106), and periodontitis (n=106). Information regarding participants' coffee consumption habits and their daily coffee intake will be collected. Clinical parameters to be measured will include plaque index, gingival index, bleeding on probing, gingival recession, and clinical attachment level.

The frequency of coffee consumption will be evaluated as daily, 1-2 times per week, 3-4 times per week, once per month, twice per month, and once per year. The amount of coffee consumed at a single occasion (cup, glass, mug, etc.) will also be recorded. In caffeinated coffee consumption, the preference for weak, moderate, or strong coffee, as well as consumption with milk, condensed milk, sugar, honey, or sweeteners will be assessed. For Turkish coffee, the consumption pattern will be categorized as unsweetened, moderately sweetened, or sweetened.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals were between 18 and 65 years

Exclusion Criteria:

* Individuals were excluded if they had smoked more than 100 cigarettes in their lifetime, were current smokers, had a diagnosis of uncontrolled diabetes mellitus, were pregnant, or were breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with periodontitis, gingivitis, and periodontal disease
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
periodontal pocket depth | Baseline
  physical methods to measure the distance from the bottom of a pocket to a reference line, usually the gingival margin or the cemento-enamel junction.
bleeding on probing | baseline
  To test for bleeding after probing, the probe is carefully introduced to the bottom of the pocket and gently moved laterally along the pocket wall. + is maximum and - is minimum.
Frequency of consumption of fermented foods | baseline
  the frequency of fermented foods is measured. The foods questioned were evaluated using a 7-point Likert-type frequency form (every day, 3-4 per week, 1-2 per week, 2 per month, 1 per month, never). In addition, the amounts of foods consumed each time were recorded, and the daily consumption amounts were obtained by dividing them by the frequency of consumption.

SECONDARY OUTCOMES:
plaque index | baseline
  an index for estimating the status of oral hygiene by measuring dental plaque that occurs in the areas adjacent to the gingival margin. 0 is minimum and 3 is maximum. The situation worsens as the score increases.
gingival index | baseline
  The Gingival Index (GI) scores each site on a 0 to 3 scale, with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding. 0 is minimum and 3 is maximum. The situation worsens as the score increases.
clinical attachment level | baseline
  The clinical attachment level (CAL) and radiographically assessed bone levels are used to assess the loss of periodontal tissue support in periodontitis, a chronic, multifactorial inflammatory disease of the periodontium.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided